CLINICAL TRIAL: NCT05017584
Title: Determining the ED90 for Intrathecal 0.75% Hyperbaric Bupivacaine for Bilateral Tubal Ligation
Brief Title: ED90 of 0.75% Bupivacaine for Bilateral Tubal Ligation (BTL)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00109119
Record Dates: First submitted 2021-08-03; First posted 2021-08-24 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Pain
Keywords: Tubal ligation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Hyperbaric bupivacaine 10.5mg (Experimental)
  Interventions: Drug: Hyperbaric bupivacaine
- Hyperbaric bupivacaine 12mg (Experimental)
  Interventions: Drug: Hyperbaric bupivacaine
- Hyperbaric bupivacaine 13.5mg (Experimental)
  Interventions: Drug: Hyperbaric bupivacaine
- Hyperbaric bupivacaine 15mg (Experimental)
  Interventions: Drug: Hyperbaric bupivacaine

INTERVENTIONS:
Drug: Hyperbaric bupivacaine — The dose for the first subject (A#X) will be 12 mg 0.75% hyperbaric bupivacaine. Two possible outcomes will be recorded: satisfactory or unsatisfactory anesthesia which is determined by occurrence of intraoperative pain and the need for intraoperative analgesia supplementation. Satisfactory analgesia will be defined as a sensory block to the T8 dermatome and the patient shall require no further supplementation for discomfort during her procedure. Unsatisfactory analgesia will be defined as a block not achieving a T8 dermatomal level or when a patient requests additional medication for discomfort at any time during her procedure.
  The dose for the next (A#X+1) will be adjusted based on the outcome from previous subjects respectively using up-down sequential allocation method with a biased-coin design. This process will continue in similar fashion with dose adjustments for next subjects to be based on outcome from subjects immediately prior.

SUMMARY:
The purpose of this study is to determine the dose of bupivacaine that provides effective pain management in 90% (ED90) of patients undergoing bilateral tubal ligation. This will guide anesthesiologists on the most effective dose to minimize intraoperative pain during this procedure. The goal is to make women as comfortable as possible when they undergo this procedure while also minimizing the amount of time they are required to remain in the hospital afterwards for monitoring.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* American Society of Anesthesiology class II or III
* bilateral tubal ligation

Exclusion Criteria:

* patient refusal
* BMI ≥ 50 kg/m2
* American Society of Anesthesiology class IV or above
* contraindication to neuraxial anesthesia
* allergy to bupivacaine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Dose (in mg) of intrathecal 0.75% hyperbaric bupivacaine that provides effective analgesia in 90% of patients undergoing bilateral tubal ligation as measured by patient reported effectiveness. | End of study, up to 2 years

SECONDARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) during surgery | End of study, up to 2 years
  Pain rating 0-10 as outlined by the NPRS by patient during procedure, in the post-anesthesia care unit, and overall at discharge
Side effects | End of study, up to 2 years
  Incidence of side effects intra-operatively
Nausea | End of study, up to 2 years
  Presence of absence of nausea
Vomiting | End of study, up to 2 years
  Presence of absence of vomiting
Itching | End of study, up to 2 years
  Presence of absence of itching
Vasopressor use | End of study, up to 2 years
  Number of participants requiring the of vasopressors (phenylephrine and ephedrine). Indicated for blood pressure drops greater than 15% below baseline or < 100mm Hg systolic.
Patient satisfaction | End of study, up to 2 years
  Overall patient satisfaction at discharge as measured by patient report. This will be obtained using a scale of 1-5 where 1 = very unsatisfied, 2 = unsatisfied, 3 = neither unsatisfied or satisfied, 4 = satisfied, and 5 = very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Taylor, MD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No